CLINICAL TRIAL: NCT06358742
Title: Evaluation of the Effect of Zinc Citrate Trihydrate Toothpaste on the Oral Plaque Microbiome Over a 12-week Period Compared to a Toothpaste Without Zinc Citrate Trihydrate
Brief Title: Evaluation of the Effect of Zinc Citrate Trihydrate Toothpaste on the Oral Plaque Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Intertek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ORL-GUM-2787
Record Dates: First submitted 2024-04-05; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-03

CONDITIONS: Dental Plaque
Keywords: microbiome; metatranscriptomics
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Toothpaste packaged in white tubes with a study label which only differentiates products with a alphanumeric code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZCT toothpaste (Experimental): Brush with zinc citrate trihydrate toothpaste twice per day, morning and evening, for 12 weeks
  Interventions: Other: ZCT toothpaste
- Control toothpaste (Placebo Comparator): Brush with control toothpaste twice per day, morning and evening, for 12 weeks.
  Interventions: Other: Control toothpaste

INTERVENTIONS:
Other: ZCT toothpaste
  Arms: ZCT toothpaste
Other: Control toothpaste
  Arms: Control toothpaste

SUMMARY:
This study is of a double-blind, randomised, parallel group study. Subjects will be enrolled onto the study according to the inclusion/exclusion criteria. After recruitment, subjects will be given a fluoride toothpaste without gum care agents to use for the 4-week run-in period prior to the commencement of the test phase of the study. Following the run-in period, baseline supragingival plaque samples will be collected 12 hours after last brushing, from the upper and lower jaws separately. Subjects will then then randomly allocated to one of two products (zinc citrate trihydrate [ZCT] toothpaste or control toothpaste) according to the randomization. Subjects will be instructed to use the toothpaste at home, brushing twice a day for 12-weeks. Supragingival plaque samples will be collected again from the upper and lower jaws after 2, 6 and 12 weeks. Plaque samples will then undergo metataxonomic and metatranscriptomic analyses.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, parallel group study and will be conducted by an independent clinical research organisation. Subjects will be enrolled onto the study according to the inclusion/exclusion criteria. After recruitment, subjects will be given a fluoride toothpaste without gum care agents to use for the 4-week run-in period prior to the commencement of the test phase of the study. This phase of the study is to ensure that all subjects are standardized to a fluoride only toothpaste. Following the run-in period, baseline supragingival plaque samples will be collected 12 hours after last brushing, from the upper and lower jaws separately, for metataxonomic and metatranscriptomic analysis respectively. Subjects will be randomly allocated to one of two products (zinc citrate trihydrate toothpaste/control toothpaste) according to the randomization schedule generated using Proc Plan procedure in SAS 9.4 suitable for 2-group parallel design study. Subjects will be instructed to use the toothpaste at home, brushing twice a day for 12-weeks. Supragingival plaque samples will be collected again from the upper and lower jaws after 2, 6 and 12 weeks. Samples are to be collected by a single clinician across the study to ensure consistency in sample collection. (Note: The study clinician could not collect samples at week 12 because of sickness. Different clinicians collected the samples instead. Data analysis showed that the week 12 samples did not match the week 0, 2 and 6 samples [higher levels of DNA indicative of different sample collection] and hence they were excluded from the analysis).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male/female volunteers
* Aged between 18 and 65 years old
* Willing to sign an informed consent and complete a medical history questionnaire
* Have at least 20 natural teeth including 5 teeth (excluding 3rd molars) in each quadrant
* Must be available for the duration of the study

Exclusion Criteria:

* The subject is an employee of Unilever or the site conducting the study
* Subjects taking part in other oral care studies for the Sponsor or any other company
* Smokers (including eCigarettes) or those who have smoked in the preceding 12 months.
* Subjects showing unwillingness, inability or lack of motivation to carry out the study procedures
* Subjects who are pregnant or nursing
* Subjects who have used mouthwashes within the 4 weeks prior to the start of the study.
* Subjects with a Modified Gingival Index score of 3 at screening
* Diabetics
* Subjects showing signs of early or untreated caries or significant periodontal disease, which in the opinion of the Study Dentist, would affect either the scientific validity of the study or, if the subject was to participate in the study, would affect their wellbeing.
* Subjects who have full or partial dentures or any oral piercings
* Subjects who have an active oral herpetic lesion or regularly suffer with oral herpetic lesions
* Subjects who regularly use medication or food supplements (including supplements which contain Zinc) in the 4 weeks prior to the start of the study, or during the study
* Subjects who have or have had a medical or oral condition which in the opinion of the study dentist would make them unsuitable for inclusion
* Known allergies to the toothpaste ingredients or to any dental materials
* Taking a course of antimicrobial medication within 4 weeks of screening or during the study
* Long term use of anti-inflammatory and/or antihistamine drugs. Intermittent use is permitted apart from 24 hours prior to the assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

PRIMARY OUTCOMES:
Plaque microbiome | 6 weeks
  Speciation of plaque bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maclure, BDS, Principal Investigator — Intertek CRS

IPD SHARING:
Plan to Share IPD: No